CLINICAL TRIAL: NCT03496844
Title: A Pilot Study of F-18 Fluciclovine-PET/CT as A Diagnostic Tool for Bone Metastases in Patients With Hormonal Sensitive and Resistant Prostate Adenocarcinoma
Brief Title: Fluciclovine-PET/CT for Bone Metastases From Prostate Adenocarcinoma
Acronym: BoneMetPETCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Blue Earth Diagnostics (Industry); Banner University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1803340164
Record Dates: First submitted 2018-04-05; First posted 2018-04-12 (Actual); Results first posted 2022-08-09 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Prostate Adenocarcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Routine F-18 fluciclovine-PET/CT scan (No Intervention): This arm will consist of prostate cancer patients who have had an F-18 fluciclovine-PET/CT scan for routine standard of care for biochemical recurrence. These patients would be asked to participate in the study only if there is a need for a standard of care bone biopsy.
- Research F-18 fluciclovine-PET/CT scan (Active Comparator): This arm will consist of prostate cancer patients who would not ordinarily obtain an Axumin-PET scan for routine standard of care but have a need for bone biopsy. This will include patients with metastatic castrate resistant prostate cancer. For example, a patient with known lymph node recurrence of prostate cancer and suspicious finding on a bone scan would be asked to participate in the study and get a F-18 fluciclovine-PET/CT scan prior to the standard of care bone biopsy.
  Interventions: Diagnostic Test: F-18 fluciclovine-PET/CT scan

INTERVENTIONS:
Diagnostic Test: F-18 fluciclovine-PET/CT scan — PET/CT imaging with F-18 fluciclovine
  Other Names: Axumin-PET scan
  Arms: Research F-18 fluciclovine-PET/CT scan

SUMMARY:
Determine diagnostic accuracy of Axumin-PET positive bone lesion by confirmatory bone biopsy.

ELIGIBILITY:
Inclusion Criteria:

1. Male
2. Be ≥ 18 years of age
3. Diagnosed with prostate cancer
4. Be willing and able to provide informed consent
5. Be informed of the investigational nature of this study

Exclusion Criteria:

1. Having a history of severe claustrophobia
2. Weight exceeding 400lbs

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Diagnosed with prostate cancer
Enrollment: 15 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2021-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip H Kuo, MD, PhD, Principal Investigator — University of Arizona; Hani Babiker, MD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to make individual participant data available to other researchers.

RESULTS

PARTICIPANT FLOW:
Groups:
- Research F-18 Fluciclovine-PET/CT Scan: This arm will consist of prostate cancer patients who would not ordinarily obtain an Axumin-PET scan for routine standard of care but have a need for bone biopsy. This will include patients with metastatic castrate resistant prostate cancer.
  F-18 fluciclovine-PET/CT scan: PET/CT imaging with F-18 fluciclovine
Period: Overall Study
Arm/Group | Research F-18 Fluciclovine-PET/CT Scan
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Research F-18 Fluciclovine-PET/CT Scan
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Non-Hispanic | 13
  White/Hispanic | 2
Region of Enrollment [Number; unit: participants]
  United States | 15
Percentage of participants who underwent bone biopsy [Count of Participants; unit: Participants]
  with bone biopsy | 13
  no bone biospy | 2

OUTCOME MEASURES:

1. Primary Outcome: True Positive and False Positive Rates of F-18 Fluciclovine-PET/CT Findings Compared to Bone Biopsy
Description: True positive and false positive rates of positive findings in the skeleton on F-18 fluciclovine-PET/CT scan compared to gold standard pathology from bone biopsy
Time Frame: 1 year
Population: Subjects who underwent bone biopsy
Measure: Number; unit: participants
Arm/Group | Research F-18 Fluciclovine-PET/CT Scan
Number analyzed (Participants) | 13
participants
  Total participants with bone biopsy | 13
  Number of Participants with Positive Bone Biopsy on Pathology | 7
  Number of Participants with Negative Bone Biopsy on Pathology | 6

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 1 week after the PET/CT scan was completed.
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Arm/Group | Research F-18 Fluciclovine-PET/CT Scan
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

LIMITATIONS AND CAVEATS:
Due to total lack of recruitment to cohort 1 consisting of Prostate Cancer patients who have had an F-18 fluciclovine-PET/CT scan for routine standard of care for biochemical recurrence, cohort 1 was dropped from the study. All consented subjects were in cohort 2.

Data collected for subjects who underwent bone biopsy; 2 subjects were found to have non-bone sites more clinically appropriate to biopsy which resulted in less bone biopsy data to analyze.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/44/NCT03496844/Prot_SAP_000.pdf